CLINICAL TRIAL: NCT01177800
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Infliximab in the Treatment of Chinese Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study to Evaluate Safety and Efficacy of Infliximab in Chinese Participants With Moderate to Severe Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013804; REMICADEPSO3004
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Infliximab; Remicade
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab (Experimental): 5 milligram per kilogram (mg/kg) infusion (a fluid or a medicine delivered into a vein by way of a needle) of infliximab administered intravenously (into a vein) at Week 0, 2 and 6 followed by maintenance regimen of 5 mg/kg infliximab at Week 14 and 22. Placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial infusion), matched to infliximab will be given at Week 10, 12 and 16. Total duration of treatment will be 26 weeks.
  Interventions: Drug: Placebo; Drug: Infliximab
- Placebo (Experimental): Placebo infusion, matched to infliximab will be given intravenously at Week 0, 2 and 6. At Week 10, 12 and 16, participants will receive 5 mg/kg infliximab intravenously. Placebo infusion will be again given at Week 14 and 22. Total duration of treatment will be 26 weeks.
  Interventions: Drug: Placebo; Drug: Infliximab

INTERVENTIONS:
Drug: Placebo — Placebo matched to infliximab given at Weeks 10, 12 and 16 in Infliximab arm and at Weeks 0, 2 and 6 in Placebo arm
Drug: Infliximab — 5 mg/kg infusion given intravenously at Week 0,2,6 (induction treatment phase) and at Week 14 and 22 in maintenance phase in infliximab arm and at Week 12 and 16 in Placebo arm.
  Other Names: Remicade

SUMMARY:
The purpose of this study is to determine the superiority and efficacy of infliximab induction therapy in chinese participants with moderate to severe plaque-type psoriasis (scaly skin rash) compared with placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial).

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), multicenter (when more than one hospital or medical school team work on a medical research study) and placebo-controlled study of infliximab in participants with moderate to severe plaque-type psoriasis. All the eligible participants will be randomly assigned to infliximab and placebo groups. The infliximab group will receive 5 milligram per kilogram (mg/kg) infliximab infusions (a fluid or a medicine delivered into a vein by way of a needle) intravenously (into a vein) at Week 0, 2 and 6 in the induction treatment phase followed by maintenance regimen of the intervention every 8 weeks up to 26 weeks. Placebo infusions will also be given at Week 10, 12 and 16. The placebo group will receive placebo infusion at Week 0, 2, 6, 14 and 22. At Week 10, participants in placebo group will then receive infliximab induction therapy. Efficacy of the participants will primarily be evaluated by percentage of participants who achieve a Psoriasis Area and Severity Index 75 (PASI) response at Week 10. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The body weight should be less than or equal to 80 kilogram
* Participants who had a diagnosis of plaque-type psoriasis (scaly skin rash) greater than or equal to 6 months before Screening (participants with concurrent psoriatic arthritis [joint pain] may be enrolled)
* Participants who had plaque-type psoriasis covering greater than or equal to 10 percent of total body surface area, Psoriasis Area Severity Index (PASI) score greater than or equal to 12 at Screening and at the Baseline
* Participants who are candidates for systemic treatment of psoriasis
* Females of childbearing potential and all men must be using adequate birth control measures and agree to use these measures and should not become pregnant (carrying an unborn baby) or plan to become pregnant up to 6 months after receiving last infusion of study drug

Exclusion Criteria:

* Participants who have nonplaque forms of psoriasis ( for example, erythrodermic, guttate, or pustular), or have current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Participants who are pregnant, nursing or planning to become pregnant within one year while enrolled in the study
* Participants who had previous treatment with infliximab
* Participants who have received agents targeted at reducing tumour necrosis factor or any biologic treatment within the previous 3 months
* Participants who have used any investigational drug within the previous 4 weeks or 5 times the half-life of the investigational agent, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (7):
- China (7):
  - Beijing
  - Beijng
  - Dalian
  - Jinan
  - Nanjing
  - Shanghai
  - Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: 5 milligram per kilogram (mg/kg) infusion (a fluid or a medicine delivered into a vein by way of a needle) of infliximab administered intravenously (into a vein) at Week 0, 2 and 6 during induction treatment phase followed by maintenance regimen of 5 mg/kg infliximab at Week 14 and 22. Placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial infusion), matched to infliximab was given at Week 10, 12 and 16. Total duration of treatment was 26 weeks.
- Placebo: Placebo infusion, matched to infliximab was given intravenously at Week 0, 2 and 6. At Week 10, 12 and 16, participants received 5 mg/kg infliximab intravenously. Placebo infusion was again given at Week 14 and 22. Total duration of treatment was 26 weeks.
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 84 | 45
Completed | 74 | 40
Not Completed | 10 | 5
Not completed — Adverse Event | 9 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal of informed consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 84 | 45 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (12.3) | 40.1 (11.1) | 39.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 10 | 34
  Male | 60 | 35 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Greater Than Equal to 75 Percent Response in Psoriasis Area and Severity Index (PASI)
Description: The PASI score is based on the assessment of the erythema (e), induration (I), scaling (S), and the body is divided into 4 regions head, trunk, upper extremities, lower extremities. The assessment was done on 4-point scale (where, 0 = none, 1 = slight, 2 = moderate, 3 = severe, and 4 = very severe). The total possible score ranges from 0 (no disease) to 72 (maximal disease). Participants with no less than 75 percent relative Baseline improvement in the PASI scores are considered to be PASI 75 responders.
Time Frame: Week 10
Population: Intent to treat (ITT) population included all participants randomly assigned to Infliximab or placebo group.
Measure: Number; unit: percentage of participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 84 | 45
percentage of participants | 81 | 2.2
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 10
Description: The DLQI is a dermatology-specific quality of life (QOL) instrument designed to assess impact of disease on a participants QOL. It is a 10-item questionnaire that, in addition to evaluating overall, QOL can be used to assess 6 different aspects: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships and treatment. Questions scored on a 4-point Likert scale: 0 (not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual items (0-3) were added to yield a total score (0-30); higher score = greater impairment of participants QOL.
Time Frame: Baseline and Week 10
Population: ITT population included all participants randomly assigned to Infliximab or placebo group. Here 'n' included those participants who were evaluable for this measure at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 84 | 45
units on a scale
  Baseline (n= 84,45) | 14.4 (6.2) | 14.4 (6.3)
  Change at Week 10 (n= 82,44) | -8.0 (7.1) | -1.5 (5.1)
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Change at Week 10: p-value was calculated by Non parametric ANOVA by van der Waerden method; Test type: Superiority or Other; p < 0.001, Non parametric ANOVA by van der Waerden

3. Secondary Outcome: Percentage of Participants With Static Physician Global Assessment (PGA) Score Less Than Equal to 1 at Week 10
Description: The Static physician global assessment (PGA) determines psoriasis lesions overall at given time point. Overall lesions graded for I (0= no evidence of plaque elevation to 5= severe plaque elevation), E (0 = no evidence of E, hyperpigmentation may be present to 5=dusky to deep red coloration), S (0 = no evidence of S to 5 = severe; very thick tenacious scale predominates). Sum of 3 scales divided by 3 gives final PGA score. Range for final score is 0 = cleared, except for residual discoloration, 1 = minimal, 2 = mild, 3=moderate, 4= marked and 5= severe; Scores should be rounded to the nearest whole number. If total ≤1.49, score = 1; if total≥ 1.50, score = 2. Percentage of participants with static PGA score <= 1 at week 10 were reported.
Time Frame: Week 10
Population: ITT population included all participants randomly assigned to Infliximab or placebo group.
Measure: Number; unit: percentage of participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 84 | 45
percentage of participants | 88.1 | 6.7
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 26
Description: The DLQI is a dermatology-specific QOL instrument designed to assess impact of disease on a participants QOL. It is a 10-item questionnaire that, in addition to evaluating overall, QOL can be used to assess 6 different aspects: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships and treatment. Questions scored on a 4-point Likert scale: 0 (not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual items (0-3) were added to yield a total score (0-30); higher score = greater impairment of participants QOL.
Time Frame: Baseline and Week 26
Population: ITT population included all participants randomly assigned to Infliximab or placebo group. 'n' included those participants who were evaluable for this measure at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 84 | 45
units on a scale
  Baseline (n= 84,45) | 14.4 (6.2) | 14.4 (6.3)
  Change at Week 26 (n= 80,42) | -10.3 (7.8) | -9.2 (6.6)
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Change at Week 26: p-value was calculated by Non parametric ANOVA by van der Waerden method; Test type: Superiority or Other; p < 0.001, Non parametric ANOVA by van der Waerden

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: The AE is defined as any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); significant disability; congenital (occurred before birth, due to parent's genetic input) anomaly.
Time Frame: Baseline up to end of study (Week 26)
Population: Safety Population included all participants randomly assigned to infliximab or placebo group.
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 84 | 45
participants
  AEs | 59 | 29
  SAE | 4 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Week 26)
Description: It was planned to collect and report adverse events as per the initial intervention received (either "Infliximab" or "Placebo"), instead of reporting by each intervention (that is, infliximab participants while on infliximab and infliximab participants while on placebo).
Arm/Group | Infliximab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/84 | 1/45
Other Adverse Events (participants affected / at risk) | 58/84 | 28/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=84) | Placebo (N=45)
Pulmonary Tuberculosis (Infections and infestations) | 2 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Metastatic Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Liver diseases (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=84) | Placebo (N=45)
Antinuclear antibody positive (Investigations) | 10 | 3
Alanine aminotransferase increased (Investigations) | 9 | 3
White blood cell count decreased (Investigations) | 4 | 3
Double stranded DNA antibody positive (Investigations) | 4 | 1
Blood uric acid increased (Investigations) | 3 | 1
Electrocardiogram T wave abnormal (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Lipids increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 5
Nasopharyngitis (Infections and infestations) | 3 | 5
Furuncle (Infections and infestations) | 3 | 1
Folliculitis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 2 | 0
Pelvic infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 10 | 5
Chest discomfort (General disorders) | 4 | 0
Pyrexia (General disorders) | 3 | 1
Fatigue (General disorders) | 1 | 2
Influenza like illness (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Apraxia (Nervous system disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Effulgent liver fire (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less